CLINICAL TRIAL: NCT05676840
Title: Comparing the Alignment Efficiency of Three Types of Nickel-titanium Archwires. A Randomized Control Trial
Brief Title: Comparing the Alignment Efficiency of Three Types of Nickel-titanium Archwires
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ziauddin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1431019DSAOM
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Crowding of Anterior Mandibular Teeth
Keywords: Nickel Titanium; Archwires; Crowding; Alignment; Nitinol
MeSH Terms: conditions — Crowding | interventions — Orthodontics; Orthodontic Appliances, Fixed

STUDY DESIGN:
Intervention Model Description: three groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional niti arch wire group (Other): all participants in this group will be placed conventional 014 niti lower archwire.
  Interventions: Procedure: orthodontic treatment with fixed appliances
- super elastic niti archwire group (Other): all participants will be given super elastic 014 lower NiTi archwire.
  Interventions: Procedure: orthodontic treatment with fixed appliances
- thermal niti archwire group (Other): all participants will be given thermal lower 014 niti archwire.
  Interventions: Procedure: orthodontic treatment with fixed appliances

INTERVENTIONS:
Procedure: orthodontic treatment with fixed appliances — comprehensive orthodontic treatment with fixed orthodontic appliances for the correction of misaligned teeth.

SUMMARY:
To compare the alignment efficiency of conventional NiTi arch wire to Thermal and Super elastic NiTi arch wires.

DETAILED DESCRIPTION:
Method: All the participants will be recruited from Ziauddin University dental OPD, each will be provided with full information about study. An informed consent form will be signed from every patient or their guardian/parents. Patients who agree to be part of this study will be included.

Subjects will be treated by Orthodontic resident under faculty supervision. Pre-treatment mandibular crowding will be assessed on dental casts. Randomization of the three groups will be done by "Opaque envelope technique" Bonding will be done using 3M uniteck brackets. After initial bonding good quality mandibular impressions will be taken and poured to obtain dental casts. Impressions and casts will be obtained at every 4 weeks interval until the initial alignment phase is complete. At the time of bonding all lower anterior teeth will be fully engaged in the archwire. The principal researcher will tag every model with an identification code before calculating measurements.

The contact point displacements will be measured with vernier caliper using the Little's index of irregularity. All measurements will be then summed and aggregated value will represent the degree of anterior irregularities.

ELIGIBILITY:
Inclusion Criteria:

* lower anterior crowding good oral hygeine all permanent lower incisors no previous orthodontic treatment

Exclusion Criteria:

* extracted or missing lower incisors poor oral hygeine relevant medical history previous orthodontic treatment

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
comparing the alignment efficiency of three types of NiTi archwires. | 4 months
  alignment of lower anterior crowding

CONTACTS AND LOCATIONS:
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No